CLINICAL TRIAL: NCT01740297
Title: Phase 1b/2, Multicenter, Open-label Trial to Evaluate the Safety and Efficacy of Talimogene Laherparepvec and Ipilimumab Compared to Ipilimumab Alone in Subjects With Unresected, Stage IIIB-IV Melanoma
Brief Title: Ipilimumab With or Without Talimogene Laherparepvec in Unresected Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110264; 2012-000307-32 (EudraCT Number)
Record Dates: First submitted 2012-11-14; First posted 2012-12-04 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Melanoma
Keywords: melanoma; talimogene laherparepvec; ipilimumab; immunotherapy
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Phase 1b was an open-label, multicenter single-arm part of the study to evaluate safety of talimogene laherparepvec in combination with ipilimumab.
  Phase 2 was an open-label multicenter, randomized design to further assess safety and to evaluate efficacy of talimogene laherparepvec in combination with ipilimumab.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1b: Talimogene Laherparepvec + Ipilimumab (Experimental): Participants received talimogene laherparepvec at an initial dose of 10⁶ plaque-forming units (PFU)/mL injected into 1 or more skin, nodal, or subcutaneous tumors. Subsequent doses of talimogene laherparepvec at 10⁸ PFU/mL began 3 weeks after the first dose and were administered every 2 weeks until complete response (CR), all injectable tumors had disappeared, confirmed disease progression per the modified immune-related response criteria (irRC), or intolerance of study treatment, whichever occurred first. Participants also received 3 mg/kg ipilimumab administered intravenously every 3 weeks for a total of 4 infusions starting at the time of the third dose of talimogene laherparepvec (week 6).
  Interventions: Drug: Talimogene laherparepvec; Drug: Ipilimumab
- Phase 2: Ipilimumab (Active Comparator): Participants received ipilimumab 3 mg/kg intravenously every 3 weeks for a total of 4 infusions starting at week 1.
  Interventions: Drug: Ipilimumab
- Phase 2: Talimogene Laherparepvec + Ipilimumab (Experimental): Participants received talimogene laherparepvec at an initial dose of 10⁶ PFU/mL injected into 1 or more skin, nodal, or subcutaneous tumors. Subsequent doses of talimogene laherparepvec at 10⁸ PFU/mL began 3 weeks after the first dose and were administered every 2 weeks until CR, all injectable tumors had disappeared, confirmed disease progression per the modified irRC, or intolerance of study treatment, whichever occurred first. Participants also received 3 mg/kg ipilimumab intravenously every 3 weeks for a total of 4 infusions starting at the time of the third dose of talimogene laherparepvec (week 6).
  Interventions: Drug: Talimogene laherparepvec; Drug: Ipilimumab

INTERVENTIONS:
Drug: Talimogene laherparepvec — Talimogene laherparepvec administered by intratumoral injection on Day 1 of Week 1, Day 1 of Week 4, then every two weeks thereafter.
  Other Names: IMLYGIC®; OncoVEX^GM-CSF; T-VEC
  Arms: Phase 1b: Talimogene Laherparepvec + Ipilimumab; Phase 2: Talimogene Laherparepvec + Ipilimumab
Drug: Ipilimumab — Ipilimumab administered intravenously every 3 weeks for a total of 4 infusions.
  Other Names: Yervoy®

SUMMARY:
Phase 1b of the study will evaluate the safety of talimogene laherparepvec in combination with ipilimumab. Phase 2 is a randomized study that will evaluate the safety and efficacy of talimogene laherparepvec in combination with ipilimumab versus ipilumumab alone.

DETAILED DESCRIPTION:
The phase 1b part is an open-label, multicenter, single-arm study where all participants will receive talimogene laherparepvec in combination with ipilimumab.

The phase 2 part of the study is an open-label, multicenter, randomized study to further assess the safety and to evaluate the efficacy of talimogene laherparepvec in combination with ipilimumab. Participants will be randomized 1:1 to receive talimogene laherparepvec plus ipilimumab or ipilimumab alone.

Participants randomized before amendment 2 will be stratified by stage of disease (stage IIIB/C, IVM1a, and stage IVM1b vs IVM1c) and v-raf murine sarcoma viral oncogene homolog B1 (BRAF) V600E (a mutation resulting in a substitution of glutamic acid for valine at codon 600) (mutation vs mutation not present). Participants randomized after amendment 2 will be stratified by stage of disease (stage IIIB/C and IVM1a vs stage IVM1b and IVM1c) and prior therapy (treatment naïve vs previously treated with systemic anticancer immunotherapy vs previously treated with systemic anticancer treatment other than immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant melanoma.
* Stage IIIB, IIIC, IVM1a, IVM1b, or IVM1c disease that is not suitable for surgical resection
* Phase1: Treatment naïve: Must not have received any prior systemic anticancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy for unresected stage IIIB to IV melanoma.
* Phase 2:

  * Either treatment naïve or received only one line of systemic anticancer therapy if v-raf murine sarcoma viral oncogene homolog B1 (BRAF) wild-type or up to two lines of systemic anticancer therapy including one BRAF inhibitor-containing regimen if BRAF mutant. Treatments given in an adjuvant setting (eg, interferon, radiotherapy, isolated limb perfusion, or investigational agents) are not considered as prior lines of therapy. No prior talimogene laherparepvec, other oncolytic virus therapies, or tumor vaccines are allowed, even if given in the adjuvant setting.
  * Subjects treated with prior ipilimumab must have had partial response (PR), complete response (CR), or at least 6 months of stable disease followed by disease progression.
  * Subjects previously treated with anti-program death-1 (PD1) or anti-cytotoxic T-lymphocyte associated antigen 4 (CTLA-4) antibodies must not have discontinued therapy due to any treatment-related adverse events including immune-related adverse events. Prior treatment-related adverse events should also be fully resolved and not requiring treatment for at least 28 days prior to randomization.
* Measurable disease defined as one or both of the following

  * at least 1 melanoma lesion that can be accurately and serially measured in at least 2 dimensions and for which the longest diameter is ≥ 10 mm and with perpendicular diameter ≥ 5 mm as measured by contrast-enhanced or spiral computed tomography (CT) scan for visceral or nodal/soft tissue disease. Lymph nodes must measure > 15 mm in their short axis to be considered measurable by CT scan.
  * at least 1 superficial cutaneous or subcutaneous melanoma lesion that can be accurately and serially measured in at least 2 dimensions and for which the short axis is ≥ 5 mm as measured by calipers
* Injectable disease (ie, suitable for direct injection or through the use of ultrasound [US] guidance) defined as follows:

  * at least 1 injectable cutaneous, subcutaneous, or nodal melanoma lesion ≥ 5 mm in longest diameter
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematologic, hepatic, renal, and coagulation functions

Exclusion Criteria:

* Primary uveal or mucosal melanoma
* History or evidence of melanoma associated with immunodeficiency states (eg, hereditary immune deficiency, organ transplant, or leukemia)
* Phase 1b: History or evidence of central nervous system (CNS) metastases
* Phase 2: Clinically active cerebral melanoma metastases. Subjects with up to 3 cerebral metastases, and neurological performance status of 0 may be enrolled, provided that all lesions have been adequately treated with stereotactic radiation therapy, craniotomy, or Gamma knife therapy, with no evidence of progression, and have not required steroids, for at least 2 months prior to enrollment.
* History or evidence of symptomatic autoimmune disease (such as pneumonitis, glomerulonephritis, vasculitis, rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematosus, scleroderma, or other), or history of autoimmune disease that required systemic treatment (ie, use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 months prior to enrollment. Replacement therapy (eg, thyroxine for hypothyroidism, insulin for diabetes mellitus) is not considered a form of systemic treatment for autoimmune disease.
* History of or plan for splenectomy or splenic irradiation
* Active herpetic skin lesions or prior complications of herpes simplex type-1 virus (HSV-1) infection (eg, herpetic keratitis or encephalitis).
* Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use
* Known human immunodeficiency virus (HIV) disease
* Known acute or chronic hepatitis B or hepatitis C infection
* Phase 1b: Prior talimogene laherparepvec, ipilimumab, other CTLA-4 inhibitors, PD-1 inhibitors, or tumor vaccine
* Phase 2: Prior talimogene laherparepvec, other oncolytic virus therapies, or tumor vaccines
* Currently receiving or less than 28 days since ending systemic anticancer treatment for unresected stage IIIB to IV melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-02-07 (Actual); Primary Completion 2016-08-23 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- United States (27):
  - Research Site, Tucson, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Santa Rosa, California
  - Research Site, Aurora, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Morristown, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Milwaukee, Wisconsin
- France (5):
  - Research Site, Bordeaux
  - Research Site, Grenoble
  - Research Site, Lille
  - Research Site, Nantes
  - Research Site, Paris
- Germany (3):
  - Research Site, Göttingen
  - Research Site, Kiel
  - Research Site, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Chesney J, Puzanov I, Collichio F, Singh P, Milhem MM, Glaspy J, Hamid O, Ross M, Friedlander P, Garbe C, Logan TF, Hauschild A, Lebbe C, Chen L, Kim JJ, Gansert J, Andtbacka RHI, Kaufman HL. Randomized, Open-Label Phase II Study Evaluating the Efficacy and Safety of Talimogene Laherparepvec in Combination With Ipilimumab Versus Ipilimumab Alone in Patients With Advanced, Unresectable Melanoma. J Clin Oncol. 2018 Jun 10;36(17):1658-1667. doi: 10.1200/JCO.2017.73.7379. Epub 2017 Oct 5. PMID 28981385
- [Background] Puzanov I, Milhem MM, Minor D, Hamid O, Li A, Chen L, Chastain M, Gorski KS, Anderson A, Chou J, Kaufman HL, Andtbacka RH. Talimogene Laherparepvec in Combination With Ipilimumab in Previously Untreated, Unresectable Stage IIIB-IV Melanoma. J Clin Oncol. 2016 Aug 1;34(22):2619-26. doi: 10.1200/JCO.2016.67.1529. Epub 2016 Jun 13. PMID 27298410
- [Background] Chesney J, Puzanov I, Collichio F, Milhem MM, Hauschild A, Chen L, Sharma A, Garbe C, Singh P, Mehnert JM. Patterns of response with talimogene laherparepvec in combination with ipilimumab or ipilimumab alone in metastatic unresectable melanoma. Br J Cancer. 2019 Aug;121(5):417-420. doi: 10.1038/s41416-019-0530-6. Epub 2019 Jul 29. PMID 31353364
- [Background] Dummer R, Hoeller C, Gruter IP, Michielin O. Combining talimogene laherparepvec with immunotherapies in melanoma and other solid tumors. Cancer Immunol Immunother. 2017 Jun;66(6):683-695. doi: 10.1007/s00262-017-1967-1. Epub 2017 Feb 25. PMID 28238174
- [Background] Chesney JA, Puzanov I, Collichio FA, Singh P, Milhem MM, Glaspy J, Hamid O, Ross M, Friedlander P, Garbe C, Logan T, Hauschild A, Lebbe C, Joshi H, Snyder W, Mehnert JM. Talimogene laherparepvec in combination with ipilimumab versus ipilimumab alone for advanced melanoma: 5-year final analysis of a multicenter, randomized, open-label, phase II trial. J Immunother Cancer. 2023 May;11(5):e006270. doi: 10.1136/jitc-2022-006270. PMID 37142291
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 centers in the United States of America, France, and Germany.
  Participants were enrolled in Phase 1b from 07 February 2013 to 08 July 2013 and in Phase 2 from 13 August 2013 to 25 February 2016.
Pre-assignment Details: In Phase 1b all participants received talimogene laherparepvec in combination with ipilimumab. In Phase 2 participants were randomized in 1:1 ratio to receive talimogene laherparepvec plus ipilimumab or ipilimumab. Participants randomized prior to Protocol Amendment 2 were stratified by disease stage and v-raf murine sarcoma viral oncogene homolog B1 (BRAF) mutation V600E; participants randomized after Amendment 2 were stratified by disease stage and prior therapy.
Groups:
- Phase 1b: Talimogene Laherparepvec + Ipilimumab: Participants received talimogene laherparepvec at an initial dose of 10⁶ plaque-forming units (PFU)/mL injected into 1 or more skin, nodal, or subcutaneous tumors with maximum total volume of 4 mL. Subsequent doses of talimogene laherparepvec at 10⁸ PFU/mL (up to 4 mL total) began 3 weeks after the first dose and were administered every 2 weeks until complete response (CR), all injectable tumors had disappeared, confirmed disease progression per the modified immune-related response criteria (irRC), or intolerance of study treatment, whichever occurred first. Participants also received 3 mg/kg ipilimumab administered intravenously every 3 weeks for a total of 4 infusions starting at the time of the third dose of talimogene laherparepvec (week 6).
- Phase 2: Talimogene Laherparepvec + Ipilimumab: Participants received talimogene laherparepvec at an initial dose of 10⁶ PFU/mL injected into 1 or more skin, nodal, or subcutaneous tumors with a maximum total volume of 4 mL. Subsequent doses of talimogene laherparepvec at 10⁸ PFU/mL (up to 4 mL total) began 3 weeks after the first dose and were administered every 2 weeks until CR, all injectable tumors had disappeared, confirmed disease progression per the modified irRC, or intolerance of study treatment, whichever occurred first. Participants also received 3 mg/kg ipilimumab intravenously every 3 weeks for a total of 4 infusions starting at the time of the third dose of talimogene laherparepvec (week 6).
Period: Overall Study
Arm/Group | Phase 1b: Talimogene Laherparepvec + Ipilimumab | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Started | 19 | 100 | 98
Received Talimogene Laherparepvec | 19 | 0 | 95
Received Ipilimumab | 18 | 95 | 92
Completed (Completed study) | 6 | 36 | 37
Not Completed | 13 | 64 | 61
Not completed — Withdrawal by Subject | 4 | 16 | 17
Not completed — Death | 8 | 46 | 40
Not completed — Lost to Follow-up | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Talimogene Laherparepvec + Ipilimumab | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab | Total
Number analyzed (Participants) | 19 | 100 | 98 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.1) | 64.2 (13.3) | 63.6 (14.0) | 63.6 (13.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 11 | 54 | 46 | 111
  ≥ 65 years | 8 | 46 | 52 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 45 | 36 | 92
  Male | 8 | 55 | 62 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 0 | 5
  Not Hispanic or Latino | 18 | 96 | 98 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Black (or African American) | 0 | 3 | 0 | 3
  Multiple | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 18 | 92 | 97 | 207
  Other | 1 | 2 | 0 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 14 | 73 | 69 | 156
    1 (Restrictive but ambulatory) | 5 | 27 | 29 | 61
Tumor, Node, Metastasis (TNM) Disease Stage [Count of Participants; unit: Participants] — Stage IIIB: Ulcerated lesion and 1 lymph node or 2-3 nodes with micrometastasis, or any-depth lesion with no ulceration, and 1 lymph node or 2-3 nodes with macrometastasis; Stage IIIC: Ulcerated lesion and 1 lymph node with macrometastasis; 2-3 nodes with macrometastasis or ≥4 metastatic lymph nodes, matted lymph nodes, or in-transit met(s)/satellite(s); Stage IV: M1a: Spread to skin, subcutaneous tissue, or lymph nodes; normal lactate dehydrogenase (LDH) level; M1b: Spread to lungs, normal LDH; M1c: Spread to all other visceral organs, normal LDH or any distant disease with elevated LDH.
  Participants
    Stage IIIB - IVM1a | 8 | 57 | 50 | 115
    Stage IVM1b/c | 11 | 43 | 48 | 102
BRAF V600 Mutation Status [Count of Participants; unit: Participants] — Mutation status of v-raf murine sarcoma viral oncogene homolog B1 (BRAF) gene was based on a gene mutation that results in an amino acid substitution from valine (V) to glutamic acid (E) at codon 600 (V600E) and/or a substitution from valine to lysine (K) (V600K).
  Participants
    Mutation | 12 | 34 | 35 | 81
    Wild-type | 7 | 60 | 62 | 129
    Missing/Unknown | 0 | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities
Description: A DLT was defined as any toxicity related to study drug which met any of the following criteria based on Common Terminology Criteria for Adverse Events version 3.0:
  * treatment-related non-laboratory adverse events (AE) ≥ grade 4
  * ≥ grade 4 immune-mediated dermatitis
  * ≥ grade 4 immune-mediated endocrinopathy (except autoimmune thyroiditis)
  * ≥ grade 3 immune-mediated enterocolitis
  * ≥ grade 3 immune-mediated hepatitis (except grade 3 that resolved to grade 1 or baseline within 28 days of onset)
  * ≥ grade 3 immune-mediated neuropathy
  * ≥ grade 3 other immune-mediated AEs including hemolytic anemia, angiopathy, myocarditis, pericarditis, temporal arteritis, or vasculitis, autoimmune thyroiditis (except grade 3 that resolved to grade 1 or baseline within 28 days of onset), blepharitis, conjunctivitis, episcleritis, iritis, scleritis, or uveitis, pancreatitis, meningitis, arthritis or polymyalgia rheumatic, nephritis, pneumonitis, psoriasis or leukocytoclastic vasculitis.
Time Frame: The DLT evaluation period was 6 weeks from the initial administration of ipilimumab (week 6 to 12).
Population: All phase 1b participants who received ≥ 1 dose of investigational product (talimogene laherparepvec or ipilimumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 19
Participants | 0

2. Primary Outcome: Phase 2: Objective Response Rate
Description: Objective response rate is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) according to the modified immune-related response criteria (irRC) assessed by the investigator. Tumors were examined clinically and by computed tomography (CT) or magnetic resonance imaging (MRI).
  CR: Complete disappearance of all lesions and no new lesions; Any pathological lymph nodes reduced in short axis to <10 mm.
  PR: Decrease in tumor burden ≥ 50% relative to baseline. Response must have been confirmed by a repeat, consecutive assessment ≥ 4 weeks from the date first documented. Participants who did not have any follow-up tumor assessments were regarded as non-responders.
Time Frame: Tumor response was assessed every 12 weeks until disease progression; median follow-up time at the primary analysis was 57.7 weeks and 68.1 weeks in each treatment group respectively.
Population: All participants randomized in phase 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
percentage of participants | 18.0 [11.0 to 26.9] | 38.8 [29.1 to 49.2]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Superiority; p = 0.002, Chi-squared, Corrected; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.5 to 5.5] — Obtained from the unstratified logistic regression model

3. Secondary Outcome: Phase 1b: Objective Response Rate
Description: as for outcome 2
Time Frame: Tumor response was assesed every 12 weeks until disease progression; median follow-up time at the primary analysis was 148.4 weeks.
Population: All phase 1b participants who received ≥ 1 dose of investigational product (talimogene laherparepvec or ipilimumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 19
percentage of participants | 52.6 [28.9 to 75.6]

4. Secondary Outcome: Phase 2: Best Overall Response
Description: Best overall response was categorized in descending order as a complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) or unevaluable (UE) based on investigator assessment according to the modified irRC.
  CR: Complete disappearance of all lesions and no new lesions; Any pathological lymph nodes reduced in short axis to <10 mm.
  PR: Decrease in tumor burden ≥ 50% relative to baseline. PD: Increase in tumor burden ≥ 25% relative to nadir. SD: Not meeting criteria for CR or PR, in absence of PD and no earlier than 77 days after the date of enrollment/randomization.
  CR, PR and PD must have been confirmed at 2 consecutive assessment ≥ 4 weeks apart.
  Assessments occurring after the start of the first subsequent anticancer therapy or removal of a lesion were not included.
Time Frame: as for outcome 2
Population: All participants randomized in phase 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
Participants
  Complete Response (CR) | 7 | 13
  Partial Response (PR) | 11 | 25
  Stable Disease (SD) | 24 | 19
  Progressive Disease (PD) | 33 | 31
  Unevaluable (UE) | 17 | 4
  Not Done (ND) | 8 | 6

5. Secondary Outcome: Phase 2: Disease Control Rate
Description: Disease control rate (DCR) was defined as the percentage of participants with a best overall response of CR, PR or SD based on investigator assessment according to the modified irRC.
  CR: Complete disappearance of all lesions and no new lesions; any pathological lymph nodes reduced in short axis to <10 mm.
  PR: Decrease in tumor burden ≥ 50% relative to baseline. SD: Not meeting criteria for CR or PR, in absence of PD and no earlier than 77 days after the date of enrollment/randomization.
  CR and PR must have been confirmed at 2 consecutive assessments ≥ 4 weeks apart.
Time Frame: as for outcome 2
Population: All participants randomized in phase 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
percentage of participants | 42.0 [32.2 to 52.3] | 58.2 [47.8 to 68.1]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.033, Chi-squared, Corrected — P-value is descriptive; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.1 to 3.4] — Obtained from the unstratified logistic regression model

6. Secondary Outcome: Phase 2: Durable Response Rate
Description: Durable response rate (DRR) was defined as the percentage of participants with a duration of response (best response of CR or PR) per modified irRC of at least 6 months. Duration of response is the time from the first confirmed CR or PR to confirmed disease progression per the modified irRC or death, whichever occurs earlier.
Time Frame: as for outcome 2
Population: All participants randomized in phase 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
percentage of participants | 13.0 [7.1 to 21.2] | 29.6 [20.8 to 39.7]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.007, Chi-squared, Corrected — P-value is descriptive; Odds Ratio (OR) = 2.8, 95% CI 2-sided [1.4 to 5.8] — Obtained from the unstratified logistic regression model

7. Secondary Outcome: Phase 2: Time to Response
Description: Time to confirmed response (TTR) was defined as the time from randomization to the date of the first confirmed CR or PR per modified irRC criteria. Participants who did not have a confirmed CR or PR were censored at their last evaluable tumor assessment date.
Time Frame: as for outcome 2
Population: All participants randomized in phase 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
months | NA [NA to NA] — Could not be estimated due to the low number of events | 5.8 [5.4 to 10.9]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.228, Log Rank — P-value is descriptive; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.80 to 2.49] — Obtained from unstratified Cox Proportional Hazard Model

8. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response was calculated only for participants with an objective response per modified irRC and was defined as the time from first confirmed objective response (CR or PR) to confirmed disease progression per the modified irRC or death, whichever was earlier. Responders who did not have an event of death or disease progression were censored at their last evaluable tumor assessment date.
Time Frame: as for outcome 2
Population: Participants randomized in phase 2 with a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 18 | 38
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

9. Secondary Outcome: Phase 2: Progression-free Survival
Description: Progression-free survival was measured from the date of randomization to the date of disease progression (as measured by modified irRC) or death on or before the data cutoff date, whichever occurred first. Participants who had no disease progression and did not die while on study were censored at the last disease assessment date.
Time Frame: From randomization until the primary analysis data cut-off date of 23 August 2016; median follow-up time was 57.7 weeks and 68.1 weeks in each treatment group respectively.
Population: All participants randomized in phase 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
months | 6.4 [3.2 to 16.5] | 8.2 [4.2 to 21.5]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.348, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.56 to 1.23] — Obtained from unstratified Cox Proportional Hazard Model

10. Secondary Outcome: Phase 2: Resection Rate
Description: Resection rate was defined as the percentage of participants who had surgical procedures for melanoma that resulted in a partial reduction or complete eradication of all previously unresectable cutaneous or visceral metastatic disease. Surgical procedures for melanoma with palliative intent (eg, for pain control) in the presence of disease progression were not considered resection.
Time Frame: as for outcome 9
Population: All participants randomized in phase 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
percentage of participants | 3.0 [0.6 to 8.5] | 5.1 [1.7 to 11.5]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.696, Chi-squared, Corrected

11. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause. Participants without an event were censored at the last date they were known to be alive. Participants with a vital status obtained after the data cut-off were censored at the date cut-off date.
Time Frame: as for outcome 9
Population: All participants randomized in phase 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.474, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.44 to 1.46] — Obtained from unstratified Cox Proportional Hazard Model

12. Secondary Outcome: Phase 2: Kaplan-Meier Estimate of Percentage of Participants Alive at Month 12 and 24
Description: The overall survival estimates at month 24 data were not mature as most participants had not been followed for 24 months at the time of data cutoff.
Time Frame: Months 12 and 24; The median (Q1, Q3) follow-up time from randomization to the primary analysis data cutoff date was 80.6 (58.3, 106.3) weeks.
Population: All participants randomized in phase 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
percentage of participants
  Month 12 | 81.4 [71.4 to 88.3] | 86.9 [78.1 to 92.4]
  Month 24 | 67.7 [53.3 to 78.5] | 76.6 [64.5 to 85.0]

13. Secondary Outcome: Phase 2: Progression-free Survival - Final Analysis
Description: Progression-free survival was measured from the date of randomization to the date of disease progression (as measured by modified irRC) or death, whichever occurred first. Participants who had no disease progression and did not die while on study were censored at the last disease assessment date.
Time Frame: From randomization until the end of study (09 March 2021); median follow-up time was 155 weeks in the Ipilimumab group and 214 weeks in the Talimogene Laherparepvec + Ipilimumab group.
Population: All participants randomized in phase 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
months | 6.4 [3.8 to 17.1] | 13.5 [5.2 to 25.0]
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.14, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.55 to 1.09] — Obtained from unstratified Cox Proportional Hazard Model

14. Secondary Outcome: Phase 2: Overall Survival - Final Analysis
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause. Participants without an event were censored at the last date they were known to be alive.
Time Frame: as for outcome 13
Population: All participants randomized in phase 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
months | 50.1 [32.0 to NA] — Could not be estimated due to the low number of events | 84.9 [41.0 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Phase 2: Ipilimumab vs Phase 2: Talimogene Laherparepvec + Ipilimumab; Test type: Other; p = 0.37, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.56 to 1.24] — Obtained from unstratified Cox Proportional Hazard Model

15. Secondary Outcome: Phase 2: Kaplan-Meier Estimate of Percentage of Participants Alive at Month 12 and 24 - Final Analysis
Time Frame: Months 12 and 24
Population: All participants randomized in phase 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 100 | 98
percentage of participants
  Month 12 | 79.9 [70.4 to 86.7] | 83.3 [74.2 to 89.4]
  Month 24 | 69.3 [58.9 to 77.5] | 72.7 [62.5 to 80.5]

16. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, where grade 1 = mild AE, grade 2 = moderate AE, grade 3 = severe AE, grade 4 = life-threatening or disabling AE and grade 5 = death related to AE.
  The investigator assessed whether each AE was possibly related to talimogene laherparepvec (T-VEC) and/or ipilimumab (Ipi).
Time Frame: From first dose of study drug to 30 days after last dose of T-VEC or 60 days after last dose of Ipi, whichever was later; median duration of treatment was 14.7 weeks in Phase 1b T-VEC + Ipi, 9.1 weeks in Phase 2 Ipi, and 21.1 weeks in Phase 2 T-VEC + Ipi.
Population: All participants who received ≥ 1 dose of investigational product (talimogene laherparepvec or ipilimumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Ipilimumab | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
Number analyzed (Participants) | 19 | 95 | 95
Participants
  All adverse events | 19 | 90 | 92
  Adverse events ≥ grade 2 | 17 | 72 | 80
  Adverse events ≥ grade 3 | 7 | 41 | 44
  Adverse events ≥ grade 4 | 2 | 4 | 6
  Serious adverse events | 6 | 34 | 34
  AEs leading to discontinuation of T-VEC | 0 | NA — Participants in this group did not receive T-VEC | 6
  AEs leading to discontinuation of ipilimumab | 0 | 17 | 13
  Fatal adverse events | 1 | 1 | 5
  T-VEC-related adverse events | 17 | NA — Participants in this group did not receive T-VEC | 82
  T-VEC-related adverse events AEs ≥ grade 2 | 12 | NA — Participants in this group did not receive T-VEC | 44
  T-VEC-related adverse events AEs ≥ grade 3 | 3 | NA — Participants in this group did not receive T-VEC | 15
  T-VEC-related adverse events ≥ grade 4 | 0 | NA — Participants in this group did not receive T-VEC | 1
  T-VEC-related serious adverse events | 1 | NA — Participants in this group did not receive T-VEC | 10
  T-VEC-related AEs leading to T-VEC discontinuation | 0 | NA — Participants in this group did not receive T-VEC | 0
  Fatal T-VEC-related adverse events | 0 | NA — Participants in this group did not receive T-VEC | 0
  Ipilimumab-related adverse events | 15 | 78 | 75
  Ipilimumab-related adverse events ≥ grade 2 | 8 | 50 | 48
  Ipilimumab-related adverse events ≥ grade 3 | 4 | 21 | 19
  Ipilimumab-related adverse events ≥ grade 4 | 1 | 2 | 1
  Ipilimumab-related serious adverse events | 4 | 19 | 14
  Ipi-related AEs leading to Ipi discontinuation | 0 | 12 | 11
  Fatal ipilimumab-related adverse events | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization until the end of study (09 March 2021); median follow-up time was 271 weeks in Phase 1, 155 weeks in the Phase 2 Ipilimumab group and 214 weeks in the Phase 2 T-VEC + Ipilimumab group. AEs are reported from first dose of study drug until 30 days after last dose of talimogene laherparepvec or 60 days after last dose of ipilimumab, whichever was later; median duration of treatment was 14.7, 9.1, and 21.1 weeks in each treatment group respectively.
Description: All-cause mortality is reported for all enrolled (Phase 1b) or randomized (Phase 2) participants.
  Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug (talimogene laherparepvec or ipilimumab).
Arm/Group | Phase 1b: Talimogene Laherparepvec + Ipilimumab | Phase 2: Ipilimumab | Phase 2: Talimogene Laherparepvec + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 9/19 | 52/100 | 45/98
Serious Adverse Events (participants affected / at risk) | 6/19 | 34/95 | 34/95
Other Adverse Events (participants affected / at risk) | 19/19 | 85/95 | 91/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Talimogene Laherparepvec + Ipilimumab (N=19) | Phase 2: Ipilimumab (N=95) | Phase 2: Talimogene Laherparepvec + Ipilimumab (N=95)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 1 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 1 | 2
Exophthalmos (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Autoimmune colitis (Gastrointestinal disorders) | 0 | 3 | 3
Colitis (Gastrointestinal disorders) | 0 | 9 | 6
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 5
Injection site reaction (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Talimogene Laherparepvec + Ipilimumab (N=19) | Phase 2: Ipilimumab (N=95) | Phase 2: Talimogene Laherparepvec + Ipilimumab (N=95)
Anaemia (Blood and lymphatic system disorders) | 0 | 5 | 11
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 10
Adrenal insufficiency (Endocrine disorders) | 1 | 3 | 2
Hypothyroidism (Endocrine disorders) | 2 | 4 | 4
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 3 | 8 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 11 | 15
Constipation (Gastrointestinal disorders) | 2 | 8 | 14
Diarrhoea (Gastrointestinal disorders) | 8 | 33 | 40
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 4
Nausea (Gastrointestinal disorders) | 9 | 26 | 36
Vomiting (Gastrointestinal disorders) | 5 | 13 | 19
Application site pain (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 10 | 7
Chest pain (General disorders) | 1 | 1 | 1
Chills (General disorders) | 11 | 4 | 50
Fatigue (General disorders) | 11 | 40 | 56
Influenza like illness (General disorders) | 3 | 1 | 27
Injection site inflammation (General disorders) | 1 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 27
Injection site reaction (General disorders) | 2 | 0 | 15
Injection site swelling (General disorders) | 0 | 0 | 5
Malaise (General disorders) | 1 | 2 | 7
Oedema peripheral (General disorders) | 2 | 5 | 14
Pain (General disorders) | 3 | 4 | 11
Performance status decreased (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 1 | 3
Pyrexia (General disorders) | 11 | 9 | 36
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 4
Oral herpes (Infections and infestations) | 0 | 0 | 6
Sinusitis (Infections and infestations) | 2 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 6
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 6 | 8
Amylase increased (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 8
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 3 | 5
Lipase increased (Investigations) | 1 | 2 | 0
Weight decreased (Investigations) | 0 | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 14 | 12
Dehydration (Metabolism and nutrition disorders) | 2 | 5 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 7 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 8 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 15 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 7 | 5
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 4
Brain oedema (Nervous system disorders) | 1 | 1 | 0
Cluster headache (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 10
Headache (Nervous system disorders) | 8 | 22 | 34
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 7
Depression (Psychiatric disorders) | 0 | 2 | 5
Insomnia (Psychiatric disorders) | 0 | 16 | 10
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 6
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 35 | 39
Rash (Skin and subcutaneous tissue disorders) | 9 | 29 | 40
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 6
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 4
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Embolism (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 6
Hypertension (Vascular disorders) | 1 | 3 | 4
Colitis (Gastrointestinal disorders) | 0 | 6 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.